CLINICAL TRIAL: NCT01353053
Title: Comparison of Two Immunosuppressive Regimens in Kidney Transplant Recipients With Deceased Donors With the Aim of Preventing the Development of Fibrosis / Atrophy of Reducing the Incidence of Cytomegalovirus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Alvaro Pacheco e Silva Filho, Federal University of Sao Paolo
Other Study IDs: 056410
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Disorder of Transplanted Kidney; Cytomegalovirus Infections
Keywords: Immunosuppression; Cytomegalovirus; Renal Transplant; Atrophy/interstitial; Conversion of tacrolimus everolimus
MeSH Terms: conditions — Cytomegalovirus Infections; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tacrolimus, Everolimus: Immunosuppression is the same for all patients in the study until the period between the 3rd and 5th weeks, when patients will be randomized to initial regimen and remain or be converted to everolimus tacrolimus.

SUMMARY:
The aim of this the study is to the assess whether the graft and patient survival, rejection rates and renal graft function after the first year will not differ between both study arms. The investigators will also the evaluate the reduction in the incidence of cytomegalovirus the and improvement of renal function of the everolimus after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI below 30,
* first transplants with PRA < 30,
* no contraindication for induction Thymoglobuline,
* age 18 years or younger than 70 years.

Exclusion Criteria:

* patients with a BMI above 30
* retransplantation
* patients hypersensitized with PRA > 30
* compared with Thymoglobulina indication for induction
* age under 18 or over 70 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A randomized study of 82 patients transplanted in first transplant recipients of deceased donor and in line for kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil